CLINICAL TRIAL: NCT04920474
Title: Protocol for a Research Sample Repository for Hematopoietic Cell Transplantation, Other Cellular Therapies and Marrow Toxic Injuries
Status: Recruiting | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Other Study IDs: NMDP IRB-1991-0002
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-03

CONDITIONS: Autologous Stem Cell Transplantation; Allogeneic Stem Cell Transplantation; Cellular Therapy; Marrow Toxic Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Up to thirty milliliters (30 mL) of blood are collected from adult patients and adult donors. For pediatric patients where the collection of the full sample is medically contraindicated, as little as one milliliter (1 mL) of blood may be collected.
  In cases where donor or patient blood samples are not available, samples may consist of any material that could potentially yield testable DNA. Types may include red cell pellets, extracted DNA, dried blood on filter paper, viable cells, and any other testable material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of the Research Sample Repository is to make blood samples available for research studies related to histocompatibility and hematopoietic cell transplantation (HCT) or other cellular therapy.

Representatives of participating centers and investigators or research groups may request access to research samples contained in the Research Sample Repository for the purpose of conducting research including:

* investigating molecular explanations for histocompatibility or clinical outcomes through analysis of genomic, epigenetic, or other biomolecular data
* evaluating the factors that affect transplant or cellular therapy outcome
* studying the distribution of HLA tissue types in different populations
* studying the success of transplantation, cellular therapies or supportive care in the management of marrow toxic injuries
* performing de-linked (anonymous) research

DETAILED DESCRIPTION:
Research samples will be accepted from the following four categories:

* Hematopoietic Cell or other Cellular Therapy Donors
* Cord Blood Units
* Hematopoietic Cell Transplantation or other Cellular Therapy Recipients
* Patients with Marrow Toxic Injury

ELIGIBILITY:
Eligibility to participate in the Research Sample Repository Protocol:

Hematopoietic Cell (HC) or Other Cellular Therapy Donors

* Donors are eligible to participate in the Research Sample Repository if they have donated or are scheduled to donate HCs or cellular therapy products to an allogeneic recipient either by a marrow harvest or by apheresis. This includes adults with and without decision making capacity and children.
* All donors registered on the National Marrow Donor Program (NMDP) Registry, regardless of whether they have been requested to donate a product for a patient, are eligible to participate in the Research Sample Repository.

Cord Blood Units (CBUs)

* Testable material from CBUs (Specimens) infused at treatment centers covered under the C. W. Bill Young Transplantation Program are eligible for inclusion in the Research Sample Repository. Material may be submitted by participating treatment centers, centralized laboratories and Cord Blood Banks.

Hematopoietic Cell Transplantation or Other Cellular Therapy Recipients

* All U.S. recipients of allogeneic or autologous HC transplants or cellular therapies are eligible to participate in the Research Sample Repository. This includes adults with and without decision making capacity and children.

Patients with Marrow Toxic Injury

* Any patient who is treated for a marrow toxic injury at a center participating in the NMDP's Radiation Injury Treatment Network (RITN) is eligible to participate in the Research Sample Repository. This includes adults with and without decision-making capacity and children.
* Eligible patients may have received support care only, growth factor support, hematopoietic stem cell transplant or other appropriate medical treatment for marrow toxic injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recipients and Donors that are involved with a stem cell transplantation process
Sampling Method: Non-Probability Sample
Enrollment: 99999999 (Estimated)
Dates: Start 1991-07 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
To make blood samples available for research studies related to histocompatibility and HCT or other cellular therapy | pre-HCT (recipient) or pre-donation (donor)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Spellman, Principal Investigator — NMDP Be The Match/CIBMTR
Locations (1):
- NMDP Biorepository, New Brighton, Minnesota, United States

REFERENCES:
- See also: Research Sample Repository Protocol — https://www.cibmtr.org/DataManagement/ProtocolConsent/ResearchSamples/pages/index.aspx